CLINICAL TRIAL: NCT03938272
Title: An Open-label Single-arm Treatment Extension Study to Evaluate the Long-term Efficacy and Safety of Oxabact for Patients With Primary Hyperoxaluria Who Completed Study OC5-DB-02
Brief Title: An Extension Study to Evaluate the Long-term Efficacy and Safety of Oxabact in Patients With Primary Hyperoxaluria
Acronym: ePHex-OLE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Parent, pivotal study (OC5-DB-02) did not meet primary endpoint. No safety concerns for early termination.
Sponsor: OxThera (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OC5-OL-02
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Results first posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Hyperoxaluria, Primary
MeSH Terms: conditions — Hyperoxaluria, Primary

STUDY DESIGN:
Intervention Model Description: Open-label study in which all patients will receive Oxabact OC5
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oxabact OC5 capsules (Experimental): Oxabact OC5 - Oxalobacter formigenes Strain HC-1
  Interventions: Biological: Oxabact OC5 - Oxalobacter formigenes Strain HC-1

INTERVENTIONS:
Biological: Oxabact OC5 - Oxalobacter formigenes Strain HC-1 — Live, commensal bacteria

SUMMARY:
Open label extension study of Oxabact OC5 in patients with primary hyperoxaluria

DETAILED DESCRIPTION:
OC5-OL-02 (ePHex-OLE) is a 2 year, open-label, extension study to evaluate the long-term efficacy and safety of Oxabact OC5 for patients with primary hyperoxaluria who completed treatment in the parent double-blind, placebo-controlled study OC5-DB-02 (ePHex).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent (as applicable for the age of the subject).
2. Participation in and completion of study OC5-DB-02.
3. Subjects who had received vitamin B6 during OC5-DB-02 study should maintain a stable dose. Subjects not receiving vitamin B6 during OC5-DB-02 must be willing to refrain from initiating pyridoxine during study participation.

Exclusion Criteria:

1. Inability to swallow size 4 capsules.
2. Use of antibiotics to which O. formigenes is sensitive.
3. Current treatment with a separate ascorbic acid preparation.
4. Pregnant or lactating women (or women who are planning to become pregnant).
5. Women of childbearing potential who are not using adequate contraceptive precautions.
6. Presence of a medical condition that the Investigator considers likely to make the subject susceptible to adverse effect of study treatment or unable to follow study procedures or any condition that is likely to interfere with the study drug mechanism of action (such as abnormal GI function).
7. Participation in any interventional study of another investigational product, biologic, device, or other agent or not willing to forego other forms of investigational treatment during this study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gesa Schalk, MD, Principal Investigator — KindernierenZentrum, Bonn, Germany
Locations (8):
- Vanderbilt University Hospital, Nashville, Tennessee, United States
- Centre Hospitalier Universitaire de Liège, Liège, Belgium
- Kindernierenzentrum Bonn, Bonn, Germany
- Hospital Vall d'Hebron, Barcelona, Spain
- Tunisia (3):
  - Hédi Chaker University Hospital, Sfax
  - Sahloul University Hospital, Sousse
  - Charles Nicolle University Hospital, Tunis
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxabact OC5 Capsules; OC5 in ePHex: Oxabact OC5 - Oxalobacter formigenes Strain HC-1: Live, commensal bacteria was received in both the Core study OC-DB-02 (ePHex) and this open label extension
- Oxabact OC5 Capsules; Placebo in ePHex: Placebo in the Core study OC-DB-02; and Oxabact OC5 - Oxalobacter formigenes Strain HC-1: Live, commensal bacteria in this open label extension
Period: Overall Study
Arm/Group | Oxabact OC5 Capsules; OC5 in ePHex | Oxabact OC5 Capsules; Placebo in ePHex
Started | 11 | 11
Completed | 0 | 1
Not Completed | 11 | 10
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Study termination by sponsor | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Oxabact OC5 Capsules; OC5 in ePHex; Oxabact OC5 Capsules; Placebo in ePHex: Oxabact OC5 - Oxalobacter formigenes Strain HC-1
  Oxabact OC5 - Oxalobacter formigenes Strain HC-1: Live, commensal bacteria
- Total: Total of all reporting groups
Arm/Group | Oxabact OC5 Capsules; OC5 in ePHex | Oxabact OC5 Capsules; Placebo in ePHex | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 8 | 15
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.0 (6.9) | 17.1 (14.2) | 15.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 3 | 7 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 2 | 2
  United Kingdom | 1 | 1 | 2
  Germany | 2 | 4 | 6
  Spain | 5 | 2 | 7
  Tunisia | 3 | 1 | 4
  United States | 0 | 1 | 1
Primary hyperoxaluria diagnosis [Count of Participants; unit: Participants] — Primary Hyperoxaluria is the result of rare genetic mutations. The three main types of primary hyperoxaluria are the result of different gene deficiencies.
  Primary Hyperoxaluria Type I is the result of mutations in the AGXT gene (alanine-glyoxylate aminotransferase) Primary Hyperoxaluria Type II is the result of mutations in the GRHPR gene (glyoxylate reductase-hydroxypyruvate reductase)
  Participants
    PH Type I | 11 | 10 | 21
    PH Type II | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Kidney Function (eGFR) After 12 and 24 Months of Open-label Oxabact Treatment
Description: Change in eGFR measured as mL/min/1.73m2. Baseline values are from the period before treatment with Oxabact. For the patients treated with Oxabact in the double-blind study, baseline is prior to treatment in that study. For patients who were treated with placebo in the double-blind study, baseline values are from the extension study, which was 48 to 52 weeks in the double-blind study.
Time Frame: 104 weeks
Population: Patients with at least one efficacy measurement in the open-label period
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m2
Arm/Group | Oxabact OC5 Capsules; OC5 in ePHex | Oxabact OC5 Capsules; Placebo in ePHex
Number analyzed (Participants) | 9 | 10
mL/min/1.73 m2
  Baseline value | 74.193 (9.952) | 58.617 (20.858)
  Month 2: number analyzed (Participants) | 7 | 9
  Month 2 | -1.568 (3.129) | -1.218 (5.255)
  Month 4: number analyzed (Participants) | 7 | 6
  Month 4 | -3.246 (8.158) | -2.932 (9.889)
  Month 6: number analyzed (Participants) | 6 | 7
  Month 6 | -9.547 (14.017) | 3.083 (8.614)
  Month 8: number analyzed (Participants) | 4 | 2
  Month 8 | -9.293 (13.633) | 7.825 (4.264)
  Month 10: number analyzed (Participants) | 2 | 2
  Month 10 | 1.798 (3.312) | 4.530 (0.665)
  Month 12: number analyzed (Participants) | 5 | 5
  Month 12 | -5.840 (11.672) | -0.994 (6.778)
  Month 15: number analyzed (Participants) | 3 | 2
  Month 15 | -5.862 (8.954) | 2.190 (0.764)
  Month 18: number analyzed (Participants) | 0 | 2
  Month 18 |  | 2.785 (0.516)
  Month 21: number analyzed (Participants) | 1 | 1
  Month 21 | -12.193 | -3.340
  Month 24: number analyzed (Participants) | 0 | 1
  Month 24 |  | -7.110

2. Secondary Outcome: Change From Baseline in Plasma Oxalate Concentration
Description: as for outcome 1
Time Frame: Up to 104 weeks
Population: Patients with at least one post-baseline plasma oxalate measurement
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Oxabact OC5 Capsules; OC5 in ePHex | Oxabact OC5 Capsules; Placebo in ePHex
Number analyzed (Participants) | 9 | 10
μmol/L
  Baseline value | 15.9 (6.6) | 18.1 (7.3)
  Month 2 Change from baseline: number analyzed (Participants) | 7 | 9
  Month 2 Change from baseline | 2.1 (7.2) | 1.1 (7.0)
  Month 4 Change from baseline: number analyzed (Participants) | 7 | 6
  Month 4 Change from baseline | 4.0 (8.5) | 1.3 (6.1)
  Month 6 Change from baseline: number analyzed (Participants) | 6 | 7
  Month 6 Change from baseline | 6.1 (10.0) | 2.3 (4.8)
  Month 8 Change from baseline: number analyzed (Participants) | 4 | 2
  Month 8 Change from baseline | 13.8 (14.6) | -5.5 (0.7)
  Month 10 Change from baseline: number analyzed (Participants) | 5 | 2
  Month 10 Change from baseline | 5.4 (6.0) | -8.5 (2.1)
  Month 12 Change from baseline: number analyzed (Participants) | 5 | 5
  Month 12 Change from baseline | 14.0 (15.7) | 0.4 (5.7)
  Month 15 Change from baseline: number analyzed (Participants) | 3 | 2
  Month 15 Change from baseline | 12.3 (9.6) | 4.0 (8.5)
  Month 18 Change from baseline: number analyzed (Participants) | 0 | 2
  Month 18 Change from baseline |  | 20.5 (24.7)
  Month 21 Change from baseline: number analyzed (Participants) | 1 | 1
  Month 21 Change from baseline | -2.3 | 4.0
  Month 24 Change from baseline: number analyzed (Participants) | 0 | 1
  Month 24 Change from baseline |  | -7.0

ADVERSE EVENTS:
Time Frame: Open label extension up to 24 months of treatment
Groups:
- Oxabact OC5 Capsules; Placeob in ePHex: Oxabact OC5 - Oxalobacter formigenes Strain HC-1
  Oxabact OC5 - Oxalobacter formigenes Strain HC-1: Live, commensal bacteria
Arm/Group | Oxabact OC5 Capsules; OC5 in ePHex | Oxabact OC5 Capsules; Placeob in ePHex
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 3/11 | 1/11
Other Adverse Events (participants affected / at risk) | 7/11 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxabact OC5 Capsules; OC5 in ePHex (N=11) | Oxabact OC5 Capsules; Placeob in ePHex (N=11)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxabact OC5 Capsules; OC5 in ePHex (N=11) | Oxabact OC5 Capsules; Placeob in ePHex (N=11)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (2)
Pharyngotonsillitis (Infections and infestations) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (4)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Eosinophil count increased (Investigations) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator may not publish the results of their cohort of subjects until the full study has been submitted for publication. They may not submit for publication or present the results of this study without allowing OxThera 30 days in which to review and comment on the pre-publication manuscript. The investigator may not submit the results of the study for publication without the prior consent of OxThera, unless the review period has passed and there has been no reaction from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT03938272/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT03938272/SAP_001.pdf